CLINICAL TRIAL: NCT02735551
Title: Effectiveness of LARC Forward Contraceptive Counseling and Same Day Placement in a Community College Population: A Randomized Intervention Project
Brief Title: LARC Forward Contraceptive Counseling at MHCC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inadequate participant enrollment during recruitment period.
Sponsor: Oregon Health and Science University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Bayer (Industry); Society of Family Planning (Other)
Responsible Party: Principal Investigator, Jacqueline Lamme, Adjunct Instructor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: OHSU IRB 15715
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-10

CONDITIONS: Contraception
Keywords: LARC; IUD; Contraceptive Implant; Contraception; Community college
MeSH Terms: interventions — Long-Acting Reversible Contraception; Referral and Consultation; Prescriptions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Non-LARC Group: Short Acting Method (Active Comparator): All groups will receive the same standardized contraceptive counseling ("LARC forward counseling"). Participants who chose a short-acting hormonal method (e.g. contraceptive pills, ring, or patch) will receive a prescription to the pharmacy of their choice, as is the current practice for students who present for contraceptive services
  Interventions: Other: Prescription for Short-Acting Hormonal Contraception
- Control Group: Referral for LARC Placement (Active Comparator): All groups will receive the same standardized contraceptive counseling ("LARC forward counseling"). Randomized to referral for LARC placement to local clinic.
  Interventions: Other: Referral for Long Acting Reversible Contraception (LARC)
- LARC Group: Same Day LARC Placement (Active Comparator): All groups will receive the same standardized contraceptive counseling ("LARC forward counseling"). Randomized to same day LARC placement (intervention).
  Interventions: Drug: Long Acting Reversible Contraception (LARC)

INTERVENTIONS:
Drug: Long Acting Reversible Contraception (LARC) — Same day LARC placement (intervention) of Mirena, Skyla, Paragard, Implanon
  Arms: LARC Group: Same Day LARC Placement
Other: Referral for Long Acting Reversible Contraception (LARC) — Referral to local clinic for LARC placement of choice (Mirena, Skyla, Paragard, Implanon, etc.)
  Arms: Control Group: Referral for LARC Placement
Other: Prescription for Short-Acting Hormonal Contraception — Participants who chose a short-acting hormonal method (e.g. contraceptive pills, ring, or patch) will receive a prescription to the pharmacy of their choice
  Arms: Non-LARC Group: Short Acting Method

SUMMARY:
This prospective randomized controlled study will evaluate if Long Acting Reversible Contraceptive (LARC) forward counseling in combination with same-day LARC placement increases overall LARC uptake within a community college population compared to LARC forward counseling and referral to a secondary clinic for LARC placement. The study will be conducted at Mount Hood Community College (MHCC) in Oregon. Participants will be enrolled into three groups. All groups will receive the same standardized contraceptive counseling ("LARC forward counseling") and participants will be able to choose between a LARC method and short-acting method of birth control.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the benefit of an on-campus birth control counseling and services clinic. Currently there are no health services that provide access to birth control located on the Mount Hood Community College (MHCC) campus. We are offering a temporary 'Birth Control Resource Center' for eligible students. All forms of birth control in this study are FDA approved.

During the study participants will undergo counseling to choose the method of birth control that is right for them. This will include watching an informational video and having a discussion with study staff. If participants choose pills, the patch the ring, or a diaphragm and do not have any contraindications to this method, they will receive a prescription for this method to be filled at the pharmacy of their choice. If participants choose Depo-Provera (the shot), they will receive their first shot on the day of their visit and a prescription for repeat shots every 3 months. If participants choose to have an IUD or Implant as their method of birth control, they will be randomized to one of two groups. There is a 50% chance of having the intrauterine device (IUD) or Implant placed immediately after the counseling session and a 50% chance of receiving a list of local clinics that can place the device at a later time.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish-speaking women.
* 17-30 years of age.
* Currently enrolled in a 2-year certificate program at Mount Hood Community College.
* At risk for pregnancy (sexually active with men or anticipate becoming sexually active in the next 6 months).
* Do not desire pregnancy within the next 12 months.
* No contraindications to LARC according to the Center for Disease Control and Prevention medical eligibility criteria (CDC MEC)

Exclusion Criteria:

* Women who are not currently sexually active with men and who do not anticipate becoming sexually active with a male partner in the next 6 months.
* Women who have had a tubal ligation or other sterilization procedure.
* Women who desire pregnancy within the next 12 months.
* Women currently already using a LARC method for contraception.

Ages: 17 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2016-04; Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Lamme, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Mount Hood Community College, Gresham, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lamme J, Edelman A, Padua E, Jensen JT. Evaluation of the challenges faced in increasing contraceptive access within a community college population. Contracept Reprod Med. 2017 Oct 23;2:25. doi: 10.1186/s40834-017-0051-8. eCollection 2017. PMID 29201430

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-LARC Group: Short Acting Method | Control Group: Referral for LARC Placement | LARC Group: Same Day LARC Placement
Started | 3 | 0 | 0
Completed | 3 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Overall, 3 participants enrolled in the study. All 3 participants chose to receive short acting methods and could not be randomized to either same day LARC placement or referral for LARC placement.
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-LARC Group: Short Acting Method | Control Group: Referral for LARC Placement | LARC Group: Same Day LARC Placement | Total
Number analyzed (Participants) | 3 | 0 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 3 |  |  | 3
  >=65 years | 0 |  |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.3 (0.58) |  |  | 21.3 (0.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  |  | 3
  Male | 0 |  |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  |  | 1
  Not Hispanic or Latino | 2 |  |  | 2
  Unknown or Not Reported | 0 |  |  | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Pacific Islander | 1 |  |  | 1
  African American/Black | 0 |  |  | 0
  Caucasian/White | 1 |  |  | 1
  Latino | 1 |  |  | 1
  Mutli-racial | 0 |  |  | 0
  American Indian/Alaska Native | 0 |  |  | 0
  Unknown | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Ongoing Use and Satisfaction
Description: Proportion of Long Acting Reversible Contraception (LARC) uptake among women, by group assignment. This will be evaluated based on participants' self-reported ongoing use and satisfaction by group assignment on the 3-month questionnaire after the initial visit. 3 months following placement of LARC device, initiation of short acting method, and those in the control group, participants will complete a questionnaire in order to assess ongoing use and satisfaction of their contraceptive method. This will be measured on the 3-month questionnaire.
Time Frame: 3 months
Population: No participants enrolled in both the Control Group or the LARC Group. All 3 participants analyzed met the criteria specified for this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-LARC Group: Short Acting Method | Control Group: Referral for LARC Placement | LARC Group: Same Day LARC Placement
Number analyzed (Participants) | 3 | 0 | 0
Participants | 3 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Participants were asked during the 3-month follow up questionnaire if they had seen a healthcare provider since their first study visits because of any problems or concerns about their birth control method.
Arm/Group | Non-LARC Group: Short Acting Method | Control Group: Referral for LARC Placement | LARC Group: Same Day LARC Placement
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/51/NCT02735551/Prot_SAP_000.pdf